CLINICAL TRIAL: NCT03590223
Title: Glycosylated Hemoglobin and the Risk of Perioperative Major Cardiovascular Events in Diabetic Patients Undergoing Coronary Bypass Revascularization
Brief Title: Glycosylated Hemoglobin and Risk of Perioperative Major Cardiovascular Events in Diabetic Patients Undergoing Coronary Bypass Revascularization (HbA1c)
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-02156 (ch17berdajs)
Record Dates: First submitted 2018-07-04; First posted 2018-07-18 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Event; Coronary Artery Bypass Graft; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Coronary Bypass Revascularization — analysis of perioperative major cardiovascular events in diabetic patients

SUMMARY:
Glycosylated Hemoglobin (HbA1c) is considered as one of the best markers to assess the glycaemia treatment over a period of 3 to 4 months, and is considered as predictive marker for perioperative mortality and morbidity. The impact of the elevated HbA1c on the risk of perioperative major cardiovascular events in patients undergoing coronary bypass revascularization (by retrospective analysis of perioperative cardiovascular events and preoperative HbA1c) is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients with Diabetes mellitus undergoing coronary bypass revascularization since 2012

Exclusion Criteria:

* disapproval of use of data for research purposes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with diabetes mellitus
  * undergoing coronary bypass revascularization at the Klinik für Herzchirurgie, Universitätsspital Basel, Spitalstrasse 21, CH 4031-Basel since 2012
  * who did not disapprove of use of data for research purposes
  * statistic stratification in serum level of glycosylated hemoglobin (HbA1c) > 6.5% and </= 6.5%
Sampling Method: Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
occurence of Major adverse cardiac events | perioperative = in hospital
  myocardial infarction, cardiac related death, stroke

SECONDARY OUTCOMES:
occurence of severe renal insufficiency | perioperative = in hospital
  application of renal replacement therapy (renal dialysis)
occurence of sternal wound infection | perioperative = in hospital
  sternal wound infection
mortality | perioperative = in hospital
  death rate perioperative

CONTACTS AND LOCATIONS:
Overall Officials: Denis Berdajs, PD Dr. med, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Herzchirurgie University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Result] https://www.pulsus.com/scholarly-articles/glycosylated-hemoglobin-and-adverse-events-following-elective-coronary-bypass-revascularization-4682.html